CLINICAL TRIAL: NCT00827021
Title: Effects of the Dose of Erythropoiesis Stimulating Agents on Cardiac-cerebrovascular Outcomes Quality of Life and Costs in Hemodialysis Patients. The Clinical Evaluation of the DOSe of Erythropoietins (C.E. DOSE) Trial
Brief Title: The Clinical Evaluation of the Dose of Erythropoietins Trial
Acronym: CEDOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Giovanni FM Strippoli, MD (Other)
Responsible Party: Sponsor-Investigator, Giovanni FM Strippoli, MD, MD, Consorzio Mario Negri Sud
Organization: Consorzio Mario Negri Sud (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM6X822T; 2008-006014-20
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hematinics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESAs 1 low dose (Experimental)
  Interventions: Drug: Erythropoiesis Stimulating Agents (ESAs): epoetin alfa, beta or any other epoetin in equivalent dose.
- ESAs 2 high dose (Active Comparator)
  Interventions: Drug: Erythropoiesis Stimulating Agents (ESAs): epoetin alfa, beta or any other epoetin in equivalent dose.

INTERVENTIONS:
Drug: Erythropoiesis Stimulating Agents (ESAs): epoetin alfa, beta or any other epoetin in equivalent dose. — 4000 IU/week I.V. Until the end of the trial
  Arms: ESAs 1 low dose
Drug: Erythropoiesis Stimulating Agents (ESAs): epoetin alfa, beta or any other epoetin in equivalent dose. — 18000 IU/week I.V. Until the end of the trial
  Arms: ESAs 2 high dose

SUMMARY:
Anaemia is a risk factor for death, cardiac-cerebrovascular events and poor quality of life in patients with chronic kidney disease (CKD). Erythropoietin Stimulating Agents (ESAs) are the most used treatment option.

The purpose of this study is

1. the evaluation of biochemical markers to determine the efficacy of individual prediction of ESAs therapy
2. to determine the benefits and harms of different ESA doses therapeutic strategy for the management of anaemia of end stage kidney disease (ESKD).

DETAILED DESCRIPTION:
Phase III pragmatic, randomized-controlled trial comparing different doses of ESAs in patients with renal anaemia.

Study Sample:

Total of 900 participants from Italy

Background and Rationale:

Anaemia is a risk factor for death, cardiac-cerebrovascular events and poor quality of life in patients with chronic kidney disease (CKD). Erythropoietin Stimulating Agents (ESA) are the most used treatment option. In observational studies higher haemoglobin (Hb) levels (around 10-13 g/dL) are associated with improved survival and quality of life compared to lower Hb levels (around 9 g/dL). Randomized studies have found that higher Hb targets, achieved and maintained with ESA, cause an increased risk of death, mainly due to adverse cardiac-cerebrovascular outcomes. It is possible that such effect is mediated by ESA dose. This hypothesis has not been formally tested and is the aim of the Clinical Evaluation of the DOSe of Erythropoietins (CEDOSE) trial.

CEDOSE is the first independent multicentre trial exploring the benefits and harms of different ESA doses therapeutic strategy for the management of anaemia of end stage kidney disease (ESKD).

Hypothesis:

ESA resistance is associated with adverse vascular outcomes and poor quality of life in ESKD.

The CEDOSE trial will evaluate the biochemical markers to determine the efficacy of individual prediction of ESAs therapy; moreover it will evaluate the benefits and harms of two fixed ESA doses and explore the role of two treatment strategies, one based on a low and one based on a high ESA dose.

Interventions and Comparison:

Patients will be randomized 1:1 to 4000 IU/week iv. versus 18000 IU/week iv. of epoetin alfa, beta or any other epoetin in equivalent doses.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18,
* End stage kidney disease and anemia
* Treatment with hemodialysis for renal replacement therapy
* no contraindications to erythropoietin stimulating agents (ESAs) or already treated with ESAs

Exclusion Criteria:

* Patients with Hb levels > 10 g/dl without ESAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
TSAT (transferrin saturation), serum albumin, serum ferritin, serum transferrin, serum C reactive protein | after randomization at month 1, 2, 3, 6, 12

SECONDARY OUTCOMES:
Cardiovascular mortality | after randomization at month 1, 2, 3, 6, 12
sudden death | after randomization at month 1, 2, 3, 6, 12
Stroke | after randomization at month 1, 2, 3, 6, 12
myocardial infarction | after randomization at month 1, 2, 3, 6, 12
hospitalizations due to acute coronary syndrome, transitory ischemic attacks, not planned coronary revascularization, peripheric revascularization. | after randomization at month 1, 2, 3, 6, 12
Thrombosis of the cardiovascular access | after randomization at month 1, 2, 3, 6, 12
Seizures | after randomization at month 1, 2, 3, 6, 12
Hypertensive events | after randomization at month 1, 2, 3, 6, 12
Quality of life (QoL) | at randomization and at 6 and 12 months
composite of all-cause mortality, non fatal myocardial infarction and stroke, hospitalizations due to acute coronary syndrome, transitory ischaemic attacks, not planned coronary revascularization procedures, peripheric revascularization procedures. | after randomization at month 1, 2, 3, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni FM Strippoli, MD, Study Chair — Fondazione Mario Negri Sud
Locations (41):
- Italy (41):
  - Ospedale Beato Angelo, Acri
  - Ospedale S. Giovanni Di Dio, Agrigento
  - Ospedale Civile di Alghero ASL n°1, Alghero
  - Ospedali Riuniti di Anzio e Nettuno, Anzio
  - Ospedale Bellaria, Bellaria
  - Policlinico S. Orsola - Malpighi, Bologna
  - "A. Perrino" Hospital, Brindisi
  - Ospedale Maggiore di Chieri ASL TO 5, Chieri
  - Ospedale Sant'Anna, San Fermo Battaglia, Como
  - Ospedale Nuovo Sant'Anna, Ferrara
  - Azienda Ospedaliera Universitaria OO.RR Foggia, Foggia
  - P.O. SUD - Formia ASL Latina, Formia
  - Ospedale S. Giovanni di Dio di Gorizia, Gorizia
  - Jesi (Carlo Urbani), Iesi
  - Centro Dialitico Diaverum, Ladispoli, Ladispoli
  - Ospedale Renzetti ASL Lanciano Vasto, Lanciano
  - Azienda ospedaliera Ospedale Civile di Legnano, Legnano
  - Ospedale Fornaroli, Magenta
  - Ospedale di Manduria, Manduria
  - Centro Dialitico Diaverum Marsala, Marsala
  - Ospedale Valle D'Itria ASL TA, Martina Franca
  - Ospedale di Nicosia, Nicosia
  - Ospedale San Giacomo, Novi Ligure
  - Ospedale G. Bernabeo, Ortona
  - Arnas Civico Di Cristina, Palermo
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Centro di Emodialisi ausl Parma, Parma
  - Ospedale S. Maria degli Angeli, Pordenone
  - P.P.I. Priverno, Priverno
  - Arcispedale S. Maria Nuova, Reggio Emilia, Reggio Emilia
  - Centro Dialitico Diaverum, Riesi, Riesi
  - Ospedale S. Barbara, Rogliano
  - Ospedale S. Eugenio ASL RMC, Roma
  - Istituto Clinico Humanitas, Rozzano, Rozzano
  - Policlinico San Donato, San Donato Milanese
  - Ospedale SS Annunziata, Sassari
  - Ospedale A.Landolfi, Solofra
  - Ospedale Alfredo Fiorini di Terracina, Terracina
  - Azienda Ospedaliera C.T.O./C.R.F./ M. Adelaide, Torino
  - Ospedale San Giovanni Bosco, Torino
  - S. Pio da Pietrelcina, Vasto

REFERENCES:
- [Background] Strippoli GF; Clinical Evaluation of the DOse of Erythropoietins Study Group (C.E. DOSE). Effects of the dose of erythropoiesis stimulating agents on cardiovascular events, quality of life, and health-related costs in hemodialysis patients: the clinical evaluation of the dose of erythropoietins (C.E. DOSE) trial protocol. Trials. 2010 Jun 9;11:70. doi: 10.1186/1745-6215-11-70. PMID 20534124
- [Derived] Saglimbene V, D'Alonzo D, Ruospo M, Vecchio M, Natale P, Gargano L, Nicolucci A, Pellegrini F, Craig JC, Triolo G, Procaccini DA, Santoro A, Di Giulio S, La Rosa S, Murgo A, Di Toro Mammarella R, Sambati M, D'Ambrosio N, Greco V, Giannoccaro G, Flammini A, Boccia E, Montalto G, Pagano S, Amaru S, Fici M, Lumaga GB, Mancini E, Veronesi M, Patregnani L, Querques M, Schiavone P, Chimienti S, Palumbo R, Di Franco D, Della Volpe M, Gori E, Salomone M, Iacono A, Moscoloni M, Treglia A, Casu D, Piras AM, Di Silva A, Mandreoli M, Lopez A, Quarello F, Catizone L, Russo G, Forcellini S, Maccarone M, Catucci G, Di Paolo B, Stingone A, D'Angelo B, Guastoni C, Pasquali S, Minoretti C, Bellasi A, Boscutti G, Martone M, David S, Schito F, Urban L, Di Iorio B, Caruso F, Mazzoni A, Musacchio R, Andreoli D, Cossu M, Li Cavoli G, Cornacchiari M, Granata A, Clementi A, Giordano R, Guastoni C, Barzaghi W, Valentini M, Hegbrant J, Tognoni G, Strippoli GF. [Effects of dose of erythropoiesis stimulating agents on cardiovascular outcomes, quality of life and costs of haemodialysis. the clinical evaluation of the DOSe of erythropoietins (C.E. DOSE) Trial]. G Ital Nefrol. 2013 Mar-Apr;30(2):gin/30.2.21. Italian. PMID 23832463